CLINICAL TRIAL: NCT04134702
Title: Acupuncture vs. Standard Therapy for Treatment of Postoperative Pain in Patients Scheduled for Arthroscopic Knee Surgery - a Pilot Non-randomized Controlled Trial
Brief Title: Acupuncture for Pain Control After Ambulatory Knee Arthroscopy
Acronym: AcuK-Scope
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BB 079/18
Record Dates: First submitted 2019-10-18; First posted 2019-10-22 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Postoperative Pain; Knee Arthroscopy; Acupuncture
MeSH Terms: conditions — Pain, Postoperative | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental): 30 patients will receive acupuncture additionally to standard pharmacological therapy of postoperative pain
  Interventions: Other: Acupuncture
- No intervention (No Intervention): 30 patients will receive just standard pharmacological therapy of postoperative pain

INTERVENTIONS:
Other: Acupuncture — Acupuncture and ear acupuncture using indwelling fixed needles, that will remained in situ several days after surgery until the patients will experience pain
  Arms: Acupuncture

SUMMARY:
Aim of the study: To investigate whether acupuncture with indwelling fixed needles reduces pain and analgesic requirement and foster mobilization in patients after arthroscopic knee surgery (AKS) Design: Prospective pilot investigation with non-randomized arm Number of patients: N = 60 (30 patients with acupuncture additional to standard pain treatment (SPT) vs. 30 patients with SPT only Inclusion criteria: Adult patients scheduled to elective AKS in general anaesthesia with < 80 min. duration Without previous opioid and psychotropic medication Given informed consentOutcome measures: Postoperative analgesic requirement; Pain intensity; Incidence of side effects; Physiological parameters; Mobilization score

ELIGIBILITY:
Inclusion Criteria:

1. Patients with an American Society of Anesthesiologists physical status of I to II scheduled for elective ambulatory arthroscopic knee surgery under standardized general anesthesia
2. Surgery time does not exceed 80 minutes
3. Patients without previous opioid and psychotropic medication
4. Patients aged between 19 and 55 years, able to fill in the study questionnaire (Appendix F)
5. Patients who have given written informed consent

Exclusion Criteria:

1. Current psychiatric disease
2. Local skin infection at the sites of acupuncture
3. Aged < 19 or > 55 years
4. Failure to follow the standardized schema of general anaesthesia
5. Surgery time more than 80 minutes
6. Intraoperative complications (bleeding, required blood transfusion more than 6 units of packed cells, cardiovascular instability, required catecholamines)
7. Patients who consumed opioid medication at least 6 months before surgery
8. Patients who are unable to understand the consent form or to fill in the study questionnaire.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Analgesic requirement | 10 days
  Total dose of ibuprofen taken by the patient during 10 days after arthroscopic knee surgery

SECONDARY OUTCOMES:
Pain intensity: verbal rating scale | 10 days after surgery
  Pain intensity measured using verbal rating scale from 0=no pain to 10=maximal pain
Side affects | 10 days after surgery
  Incidence of analgesic induced side effects

CONTACTS AND LOCATIONS:
Overall Officials: Taras Usichenko, MD, PhD, Study Chair — Dept. of Anesthesiology
Locations (1):
- University Medicine of Greifswald, Greifswald, Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: Yes
On request from study chair after publication of results
Supporting Information: Study Protocol, SAP, ICF, CSR